CLINICAL TRIAL: NCT03737825
Title: Computerized Cognitive Training for Patients With Cognitive Deficits Due to Multiple Sclerosis: a Pilot Study
Brief Title: Computerized Cognitive Training in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-25685
Record Dates: First submitted 2018-11-06; First posted 2018-11-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Cognitive Decline
Keywords: MS; Multiple Sclerosis; Cognitive remediation; Brain training; Physical Therapy
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking: Triple (Participant, Investigator, Outcomes Assessor) Study assessment administrator is blinded to what digital tool the subject has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Program 1 (Active Comparator): Computerized gaming rehabilitation Program 1.
  Interventions: Device: Computerized gaming rehabilitation Program 1
- Program 2 (Placebo Comparator): Computerized gaming rehabilitation Program 2.
  Interventions: Device: Computerized gaming rehabilitation Program 2

INTERVENTIONS:
Device: Computerized gaming rehabilitation Program 1 — Brain training games displayed on a large screen paired with physical exercise component. The program involves movements such as reaching, stepping, or stretching in place.
  Arms: Program 1
Device: Computerized gaming rehabilitation Program 2 — Brain training games displayed on a tablet device paired with physical exercise component. The program involves movements such as reaching, stepping, or stretching.
  Arms: Program 2

SUMMARY:
WHO: 40 participants with a confirmed diagnosis of Multiple Sclerosis (MS) able to engage in moderate physical activity.

WHY: The purpose of this study is to evaluate two computerized brain training tools, which include light physical activity, to see if they can help improve cognitive functions, such as memory and attention, for patients with MS.

WHAT: Complete a set of tests (physical and cognitive) at baseline, wear a Fitbit Flex device at home for the duration of the study, 3 supervised sessions for 4 weeks at UCSF, one visit for physical and cognitive tests at one week after the final supervised session, and one final visit 6 months after the final supervised session.

WHERE: 20 participants at the UCSF Weill Institute for Neurosciences (675 Nelson Rising Lane, San Francisco, CA); 20 participants at Lausanne University Hospital (Rue du Bugnon 46, 1005 Lausanne, Switzerland)

DETAILED DESCRIPTION:
This is a dual-site trial with identical study activities taking place at both locations. If you live in/near San Francisco, study visits will take place at UCSF; if you live in/near Lausanne, Switzerland, study visits will take place at the Lausanne University Hospital.

You will be asked to attend one initial session for cognitive tests and answer questions regarding your medical history to see if you are eligible for the study. This process takes about 20 minutes. If you are eligible you will be asked to schedule the following appointments to participate:

First you will be randomized into one of two different training programs. You will not be able to choose which program you are placed in, but have equal chances of being randomized into each:

* Program 1 involves brain training games displayed on a large screen. Participants will use whole-body movements to complete game tasks. Tasks involve movements such as reaching, stepping, and jogging in place. These movements are tracked by a motion sensor. Stretching, warm-up, and cool down sessions will be mandated prior to and following the tasks.
* Program 2 involves brain training and guided, light physical exercise games on a tablet device. The exercise involves movements such as reaching, stepping, and stretching. Stretching, warm-up, and cool down sessions will be mandated prior to and following the tasks.

Baseline Visit: This session should take about two hours. You will be given some cognitive, visual and physical tests. You will be given questionnaires about your mood, fatigue and function. You will receive a Fitbit Flex to be worn daily for the duration of the study. The Fitbit will track daily active step count, number of active minutes, quality/length of sleep cycles.

Week 1-4 Visits (12 sessions in total): These sessions will be 1 hour and 30 minutes each (Note: the first session will be 2 hours to account for calibrations). You will come in three times a week for four weeks to attend on-site sessions. You will be asked to complete digital, cognitive and physical training at each one of these visits.

Post-Training Visit: You will be asked to come in for an assessment 1 week after completing your last training session. This visit will take about 2 hours. You will be asked to complete some cognitive, visual, and physical tests. You will be given questionnaires on mood, fatigue, and everyday function. You will also return the Fitbit you received at the start of the study.

A final follow-up visit will occur 6 months after you have completed your last training session. This visit will take about two hours. You will be asked to complete some cognitive, visual and physical tests. You will be given questionnaires on mood, fatigue and function.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Presence of subjective cognitive complain from patient
* Objective general cognitive impairment: paper-and-pencil Symbol Digit Modalities Test (SDMT) z-score < -0.5 at screening

Exclusion Criteria:

* Falls in the past 12 weeks as evaluated in the enrollment interview [Hopkins Falls Grading Scale (Grade >1)]
* Strong risk of falling, assessed using the miniBEST (score< 16)
* Psychiatric co-morbidity or anti-depressive or anxiolytic medication that has been changed over the 6 months preceding consideration for study enrollment
* Colorblindness
* Presence of clinically and/or radiologically confirmed relapses or disease progression in the past 12 weeks.
* Visual, mental, motor or brainstem Functional Systems Score (FSS) on the Expanded Disability Status Scale (EDSS) superior to 2.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Change in processing speed after 4 weeks of treatment with computerized gaming rehabilitation paired with physical activity 'Program 1', vs. 'Program 2'. | 4 weeks
  Processing speed is being measured by the Symbol Digit Modalities Test (SDMT) score. SDMT measures the time to pair abstract symbols with specific numbers. The test requires visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items in 90 seconds. (max=110, min=0). Higher scores indicate improvement. Lower scores indicate worsening.

SECONDARY OUTCOMES:
Change in attention after 4 weeks of treatment with computerized gaming rehabilitation paired with physical activity 'Program 1', vs. 'Program 2'. | 4 weeks
  Attention is measured by the Test of Variables of Attention (TOVA). This computerized culture- and language-free test uses both visual and auditory stimuli to assess the speed and accuracy of attentional processing deficits in the domain of attention (Greenberg, 1998). Initially devised for ADHD in children, its predictive power has been demonstrated in other patient groups with attention and memory impairments (Braverman et al., 2006): domains also largely impaired in MS. The TOVA has furthermore been chosen here because positive effects following BBT training in young adults have been observed on this test (ongoing study at the Neuroscape Center at UCSF, unpublished data).
Change in visual working memory after 4 weeks of computerized gaming rehabilitation paired with physical activity 'Program 1', vs. 'Program 2'. | 4 weeks
  Visual working memory will be assessed via performance on 'Filter task', an established assessment of visual working memory Vogel, McCollough, & Machizawa, 2005).
Change in multitasking performance following 4 weeks of computerized paired with physical activity 'Program 1', vs. 'Program 2'. | 4 weeks
  The Triangle Tracer module of ACE evaluates multitasking abilities and is based on the same principles as Neuroracer, UCSF Neuroscape's paradigm for assessment and training of multitasking (Anguera et al., 2013)
Change in working memory following 4 weeks of computerized paired with physical activity 'Program 1', vs. 'Program 2'. | 4 weeks
  The Brief Visuospatial Memory Test (BVMT) is an immediate non-verbal recall test, and a standardized assessment tool of working memory in MS.

OTHER OUTCOMES:
Change in mood after 4 weeks treatment with Program 1 vs. Program 2. | 4 weeks
  Mood is measured by the Center for Epidemiological Studies - Depression (CES-D), which asks participants to rank 20 different symptoms on a severity scale of 0 to 3. The score is the sum of these subscales (max=60, min=0). Scores of 16 or greater are indicative of higher risk for clinical depression.
Change in fatigue after 4 weeks treatment with Program 1 vs. Program 2. | 4 weeks
  Fatigue is being measured by the Modified Fatigue Impact Scale (MFIS) which has participants rank 21 items on 0 to 4 (never to always) scale. The score is the sum of these subscales. (max=84, min=0) Lower scores indicate improvement. Higher scores indicate worsening.
Improvement in MS-related outcomes after 4 weeks treatment with Program 1 vs. Program 2. | 4 weeks
  These outcomes will include MSQOL54 that has patients rank responses to 12 sub-scales: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. This provides a composite score (min=0, max=100) which can be broken down into two summary scores for physical health and mental health. These scores are derived from a weighted combination of scale scores.
Improvement in cognition outcomes after 4 weeks treatment with Program 1 vs. Program 2. | 4 weeks
  The outcomes will include MSNQ composite score (min=0, max=60). Scores >27 indicate cognitive impairment.
Change in attentional behavior after 4 weeks of treatment with Program 1 vs Program 2. | 4 weeks
  The Rating Scale of Attentional Behavior (RSAB) is a 14-item questionnaire and validated standard assessment of everyday life attention. A higher composite score (min=0, max=75) indicates poor attentional behavior.
Change in anxiety after 4 weeks of treatment with Program 1 vs Program 2. | 4 weeks
  Both state and trait anxiety are measured by the State Trait Anxiety Inventory (STAI). The outcome is a composite score (min=20, max=80) for STAI-state and STAI-trait sub-scales. Higher scores indicate greater anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Riley Bove, MD, Principal Investigator — University of California, San Francisco; Arseny Sokolov, MD, Principal Investigator — Centre hospitalier universitaire vaudois, Lausanne
Locations (2):
- Weill Institute for Neurosciences, University of California, San Francisco, San Francisco, California, United States
- Lausanne University Hospital (CHUV), Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braverman ER, Chen TJ, Schoolfield J, Martinez-Pons M, Arcuri V, Varshavskiy M, Gordon CA, Mengucci J, Blum SH, Meshkin B, Downs BW, Blum K. Delayed P300 latency correlates with abnormal Test of Variables of Attention (TOVA) in adults and predicts early cognitive decline in a clinical setting. Adv Ther. 2006 Jul-Aug;23(4):582-600. doi: 10.1007/BF02850047. PMID 17050501
- [Background] Forbes GB. Clinical utility of the Test of Variables of Attention (TOVA) in the diagnosis of attention-deficit/hyperactivity disorder. J Clin Psychol. 1998 Jun;54(4):461-76. doi: 10.1002/(sici)1097-4679(199806)54:43.0.co;2-q. PMID 9623751
- [Background] Anguera JA, Boccanfuso J, Rintoul JL, Al-Hashimi O, Faraji F, Janowich J, Kong E, Larraburo Y, Rolle C, Johnston E, Gazzaley A. Video game training enhances cognitive control in older adults. Nature. 2013 Sep 5;501(7465):97-101. doi: 10.1038/nature12486. PMID 24005416
- [Background] Vogel EK, McCollough AW, Machizawa MG. Neural measures reveal individual differences in controlling access to working memory. Nature. 2005 Nov 24;438(7067):500-3. doi: 10.1038/nature04171. PMID 16306992